CLINICAL TRIAL: NCT05740644
Title: Clinical Evaluation of the Zynex Monitoring System, Model CM-1600
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zynex Monitoring Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PR 2022-516
Record Dates: First submitted 2023-02-13; First posted 2023-02-23 (Actual); Results first posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-06

CONDITIONS: Fluid Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Blood Loss and Saline Infusion (Experimental)
  Interventions: Device: CM-1600

INTERVENTIONS:
Device: CM-1600 — Healthy subjects undergoing a manual blood loss of up to 500mL followed by an infusion of 1 liter of normal saline will be connected to the CM-1600 device.

SUMMARY:
This is a prospective, single-arm, non-randomized, non-controlled single-center study for the evaluation of the Zynex CM-1600 in 20 healthy adults undergoing a manual blood loss of up to 500mL followed by an infusion of 1 liter of normal saline.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have the ability to understand the parameters of participation and provide written informed consent
* Male or female of any race
* Participant is adult 18 or older
* Participant must be willing and able to comply with study procedures and duration
* In the Principal Investigator's medical judgment, the participant is suitable for a blood draw of up to 500mL
* Participant must weigh at least 110 pounds

Exclusion Criteria:

* Any upper extremity amputation
* Females who are pregnant, who are trying to get pregnant, or have a urine test positive for pregnancy on the day of the study
* Participant has a heart condition that may interfere with the Zynex CM-1600 (e.g., pacemakers, defibrillator, irregular heartbeat, dextrocardia, etc.)
* Participant has been diagnosed with chronic fatigue syndrome (also known as chronic fatigue, immune dysfunction syndrome, or myalgic encephalomyelitis)
* Participant requires equipment and/or devices that may interfere with the Zynex CM-1600 (e.g., life-sustaining equipment, other monitoring devices, insulin pumps, or other implanted devices)
* Participant is taking coumadin (warfarin), heparin, or other prescription blood thinners for 7 or more days prior to blood draw
* Participant donated blood within 8 weeks prior to the study blood draw
* Participant has high or low blood pressure on the day of blood draw (high blood pressure is defined as systolic > 180 mmHg or diastolic > 100 mmHg; low blood pressure is defined as systolic < 100 mmHg or diastolic < 60 mmHg)
* Participant has symptoms of an active infection or a temperature ≥ 100 °F
* Female with hemoglobin levels of less than 12.1g/dL or male with hemoglobin levels of less than 13.8g/dL
* Participants with self-reported heart or cardiovascular conditions such as:

  * History of cardiovascular surgery
  * History of chest pain (angina)
  * Heart rhythms other than a normal sinus rhythm or respiratory sinus arrhythmia
  * History heart attack/myocardial infarction
  * Peripheral arterial disease
  * Carotid artery disease
  * Unexplained shortness of breath
  * Congestive heart failure (CHF)
  * History of stroke/transient ischemic attack
  * Myocardial ischemia
  * Cardiomyopathy
  * Dextrocardia
* Participants with clotting disorders such as:

  * Hemophilia
  * History of blood clots
  * History of bleeding problems
  * Bruises easily
* Self-reported health conditions as identified in the Health Assessment Form including:

  * Diabetes
  * Uncontrolled thyroid disease
  * Kidney disease / chronic renal impairment
  * History of seizures (except childhood febrile seizures)
  * Epilepsy
  * History of unexplained syncope
  * Recent history of frequent migraine headache within the last 2 months
  * Recent head injury within the last 2 months
  * History of cancer, with or without chemotherapy within the last 2 months
* Other known health conditions deemed unsuitable for participation by the PI when considered upon disclosure on health assessment form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinimark, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.zynexmonitoring.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Blood Loss and Saline Infusion
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Blood Loss and Saline Infusion
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: CM-1600 Ability to Detect Minor Blood Loss
Description: The objective of this study is to determine if manual blood loss of up to 500mL of blood can be identified using the non-invasive Zynex CM-1600. This will be measured by determining the percent change in Relative Index (RI) before and after the Blood Draw. The RI is an investigational value which utilizes proprietary algorithms to combine the changes of multiple measured parameters (utilizing a weighted summation of percent change values) which are indicative of relative changes in fluid volume in adult patients into a single value. The RI is a unitless value with no set minimum or maximum, where 100 is a patient's baseline. Based on the nature of the RI itself, a direct interpretation of a positive or negative outcome cannot be derived from the absolute value, instead it could be used to monitor trending of a patient's parameters relative to their baseline.
Time Frame: Duration of Recovery Period following blood draw (10 minutes)
Measure: Mean (Standard Deviation); unit: Percent change in RI
Groups:
- Blood Loss: CM-1600: Healthy subjects undergoing a manual blood loss of up to 500mL while being connected to the CM-1600 device.
Arm/Group | Blood Loss
Number analyzed (Participants) | 20
Percent change in RI | 8.0 (23.6)

2. Primary Outcome: CM-1600 Ability to Detect Saline Reinfusion
Description: The objective of this study is to determine if a saline reinfusion of 1000mL of normal saline can be identified using the non-invasive Zynex CM-1600. This will be measured by determining the percent change in Relative Index (RI) before and after the Saline Reinfusion. The RI is an investigational value which utilizes proprietary algorithms to combine the changes of multiple measured parameters (utilizing a weighted summation of percent change values) which are indicative of relative changes in fluid volume in adult patients into a single value. The RI is a unitless value with no set minimum or maximum, where 100 is a patient's baseline. Based on the nature of the RI itself, a direct interpretation of a positive or negative outcome cannot be derived from the absolute value, instead it could be used to monitor trending of a patient's parameters relative to their baseline.
Time Frame: Recovery period following saline reinfusion (10 minutes)
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Saline Reinfusion: CM-1600: Following a manual blood loss of 500mL, healthy subjects receive an infusion of 1 liter of normal saline while being connected to the CM-1600 device.
Arm/Group | Saline Reinfusion
Number analyzed (Participants) | 20
Percent change | 10.2 (38.2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during subject participation in the study and for 24hrs following (e.g., up to 48hrs)
Arm/Group | Blood Loss and Saline Infusion
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-12): https://cdn.clinicaltrials.gov/large-docs/44/NCT05740644/Prot_SAP_000.pdf